CLINICAL TRIAL: NCT04164641
Title: Noraxon myoRESEARCH™ Software Gait Analysis Evaluation and Orthotic Gait Correction in Reducing Diabetic Foot Ulceration Or Subsequent Amputation in Patients With a History of a Diabetic Foot Ulceration
Acronym: NECRO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00208316
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: Prospective, Single Center, Non-Randomized, Single treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Noraxon myoRESEARCH™ Software (Experimental): All participants will be assigned to this group to receive study intervention.
  Interventions: Device: Noraxon myoRESEARCH™ Software Gait Analysis Evaluation and Orthotic

INTERVENTIONS:
Device: Noraxon myoRESEARCH™ Software Gait Analysis Evaluation and Orthotic — Physical therapy evaluation (range of motion, strength, mobility, scale). Noraxon based gait assessment on treadmill while barefoot and with instrumented inner soles. Over ground walking assessment (with wireless instrumented inner soles, observational gait analysis while climbing stairs, ramps, curbs). Noraxon gait assessment and walking on treadmill will be video recorded for assessment. Standard measure of functionality and 6 minute walk test will be conducted. Patient will be fitted with corrective orthotics, based on usual care. Physical therapy re-evaluation. Noraxon based gait assessment and foot assessment (any areas of irritation, callus formation, swelling, ulcer formation, and gait mobility irregularities will be monitored and reassessed) throughout the study.

SUMMARY:
Determining whether the utilization of Noraxon myoRESEARCH Software gait analysis Evaluation and orthotic gait Correction can reduce diabetic foot ulceration Or subsequent amputation in patients with a history of a diabetic foot ulceration.

DETAILED DESCRIPTION:
The purpose of this study is to identify emerging abnormal structural pathology of the vulnerable re-ulcerative diabetic foot incorporating physical therapy evaluation as well as the Noraxon gait analysis to generate quantitative and qualitative gait data. Once peak foot pressures and gait pathology is identified, gait remedy is fabricated including either a foot orthotic and/or an ankle foot prosthesis. Evaluation of constructed remedy will then be evaluated focusing on gait analysis data to validate decreased plantar foot peak pressures and gait realignment towards the reduction of the diabetic foot re-ulceration and subsequent foot or limb loss.

ELIGIBILITY:
Inclusion Criteria:

* History of healed diabetic foot ulceration
* Over 18 years of age

Exclusion Criteria:

Patients who are:

* under 18 years of age
* non-diabetic
* non-ambulatory
* non-healed wounds.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of re-ulceration occurrences | One year
  Number of re-ulceration occurrences will be assessed to determine the rate of re-ulceration in patients.

SECONDARY OUTCOMES:
Number of major proximal amputation occurrences | One year
  Number of major proximal amputation occurrences will be counted.
Change of peak plantar pressure (n/cm^2) | Every 3 months, up to one year
  Assessment will be done at follow up visits.
Change of length of gait (m) | Every 3 months, up to one year
  Assessment will be done at follow up visits.
Location of amputation | One year
  If any amputation occurs, the location (level of amputation) will be assessed by looking at the stump or from information in patient medical records. Locations include below the knee (transtibial), at the knee (knee disarticulation), above the knee (transfemoral) and at the hip (hip disarticulation).
Number of patients who remain in remission | One year
  Remission is defined as being ulcer free.
Percentage of patients who do not experience re-ulceration after custom orthosis | One year
  The percentage of patients who do not experience re-ulceration after custom orthosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Sherman, DPM, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No